CLINICAL TRIAL: NCT02478840
Title: A Single Center, Open Label Clinical Trial Investigating the Long-term Efficacy of rhLAMAN (Recombinant Human Alpha-mannosidase or Lamazym) Treatment in Subjects With Alpha-Mannosidosis Who Previously Participated in Lamazym Trials
Brief Title: Evaluation of Long-term Efficacy of Treatment With Lamazym
Acronym: rhLAMAN-10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zymenex A/S (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rhLAMAN-10
Record Dates: First submitted 2015-02-09; First posted 2015-06-23 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamazym (Experimental): 1 mg Lamazym/kg Body weight
  Interventions: Drug: Lamazym

INTERVENTIONS:
Drug: Lamazym — recombinant human alpha-mannosidase
  Other Names: rhLAMAN

SUMMARY:
The overall objective is to evaluate the long-term efficacy of Lamazym i.v. treatment in patients with alpha-Mannosidosis previously enrolled in Lamazym trials and currently receiving the treatment according to the AfterCare Program.

DETAILED DESCRIPTION:
The primary objective of the trial is to evaluate the impact of the long-term treatment with Lamazym upon the level of biomarker oligosaccharides in serum and upon the endurance as measured by the change from baseline in the number of steps climbed in 3 minutes (3MSCT).

As secondary objectives, the long term efficacy of Lamazym will be investigated upon endurance as measured by the change from baseline in the number of meters walked in six minutes (6MWT), upon pulmonary function, motor proficiency by BOT-2 and hearing capability by audiometry. In addition, cognitive development will be assessed by Leiter-R test. CNS involvement will be evaluated with MRI/MRS (for patients who previously participated in rhLAMAN-02 trial), CSF biomarkers (Tau, NFL, GFAp) and CSF biomarkers oligosaccharides. Clearance of oligosaccharides in urine will be measured.

Long-term safety and Pharmaco-Kinetic (PK) profile after long-term treatment as measured by rhLAMAN levels in plasma will be assessed as well.

Quality of life will be assessed by questionnaires (CHAQ and EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have participated in the phase 1 trial (EudraCT number: 2010-022084-36), phase 2a trial (EudraCT number: 2010-022085-26), phase 2b trial (EudraCT number: 2011-004355-40) or phase 3 trial (EudraCT number: 2012-000979-17)
2. The subject must still be receiving weekly intravenous infusions of Lamazym according to the AfterCare Program
3. The Subject or subjects legally authorized guardian(s) must provide signed, informed consent prior to performing any trial-related activities
4. The subject and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

1. History of bone marrow transplantation
2. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial. Subjects unable to perform the motor tests independently from support are permitted to participate in the trial and will be evaluated for the remnant non motor endpoints
3. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the trial
4. Pregnant and/or lactating women cannot participate in the trial. Concerning women of child bearing potential (WOCBP), the investigators will decide whether or not there is a need for contraception. This assessment will be done through interviews with the patient and parents.
5. Participation in other interventional trials testing IMP, including rhLAMAN-07 (EudraCT number: 2013-000336-97) and rhLAMAN-09 (EudraCT number: 2013-000321-31) trials with Lamazym
6. Pause of the IMP for 2 consecutive weeks during the last month. Subjects are allowed to be re-screened

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in reduction of oligosaccharides in serum | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Primary Endpoint evaluation as change
Change from baseline in 3 Minutes Stair Climb Test (3MSCT) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Primary Endpoint evaluation as change

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Pulmonary function: Forced Vital Capacity (FVC) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Pulmonary function: Forced Expiratory Volume during first second (FEV1) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Pulmonary function: Peak Expiratory Flow Rate (PEF) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Functional capacity according to Bruininks-Oseretsky test of Motor Proficiency (BOT-2) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Pure Tone Audiometry (PTA) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Equivalence age measured by Leiter International Performance Scale-Revised (Leiter-R) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Assessment of mannose-rich oligosaccharides in brain tissue as measured by Magnetic Resonance Spectroscopy (MRS) visual score (for patients who previously participated in rhLAMAN-02) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Assessment of mannose-rich oligosaccharides in brain tissue as measured by Magnetic Resonance Imaging (MRI) diffusion coefficient (for patients who previously participated in rhLAMAN-02) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Cerebrospinal fluid biomarkers: Oligosaccharides in Cerebrospinal Fluid (CSF) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Cerebrospinal fluid neuro-degeneration biomarkers: Tau Protein (Tau) in Cerebrospinal Fluid (CSF) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Cerebrospinal fluid neuro-degeneration biomarkers: Neurofilament Protein Light (NFL) in Cerebrospinal Fluid (CSF) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Cerebrospinal fluid neuro-degeneration biomarkers: Glial Fibrillary Acidic protein (GFAp) in Cerebrospinal Fluid (CSF) | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  Endpoint evaluation as change
Drug exposure by Pharmaco Kinetic (PK) sampling profile on plasma | 1 week
  Evaluation of steady state Pharmaco Kinetics
Measurement of in vivo biological activity of Lamazym in blood before and after Infusion of Lamazym | 1 week
  Comparing with Anti Body (AB) and PK measurements. Measuring unit is mU/mL
Oligosaccharides in urine | 1 week
  Evaluation of steady state

OTHER OUTCOMES:
Quality of life based on questionnaires | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  filled by the subject's guardian, will be evaluated by Childhood Health Assessment Questionnaire (CHAQ) questionnaires filled in by the subject's guardian, will be evaluated by CHAQ and EQ-5D-5L
Quality of life based on questionnaires | Baseline evaluation prior to first dose compared to evaluation after one, two or four years of treatment
  filled by the subject's guardian, will be evaluated by Health Questionnaire (EQ-5D-5L) questionnaires filled in by the subject's guardian, will be evaluated by CHAQ and EQ-5D-5L
Development of adverse events | 1 week
  Safety endpoint assessed from signing of the Informed Consent Form (ICF)
Development of clinically significant changes in vital signs and change in physical examination | 1 week
  Safety endpoint assessed throughout the trial
Development of clinically significant changes in the clinical laboratory Parameters: Hematology | 1 week
  Safety endpoint assessed throughout the trial
Development of clinically significant changes in the clinical laboratory Parameters: Biochemistry | 1 week
  Safety endpoint assessed throughout the trial
Development of clinically significant changes in the clinical laboratory Parameters: Urinalysis | 1 week
  Safety endpoint assessed throughout the trial
Development of rhLAMAN antibodies | 1 week
  Safety endpoint assessed throughout the trial
Development of rhLAMAN neutralizing/inhibitory antibodies | 1 week
  Safety endpoint assessed throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Allan M Lund, MD, Principal Investigator — Copenhagen University Hospital, Center for Metabolic Diseases, Department of Clinical Genetics; Jens M Fogh, DVM, Study Chair — Zymenex A/S
Locations (1):
- Center for Metabolic Diseases, Department of Clinical Genetics, Juliane Marie Centre, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen, Denmark

REFERENCES:
- [Background] Phillips D, Hennermann JB, Tylki-Szymanska A, Borgwardt L, Gil-Campos M, Guffon N, Amraoui Y, Geraci S, Ardigo D, Cattaneo F, Lund AM. Use of the Bruininks-Oseretsky test of motor proficiency (BOT-2) to assess efficacy of velmanase alfa as enzyme therapy for alpha-mannosidosis. Mol Genet Metab Rep. 2020 Apr 8;23:100586. doi: 10.1016/j.ymgmr.2020.100586. eCollection 2020 Jun. PMID 32292699
- [Background] Borgwardt L, Guffon N, Amraoui Y, Jones SA, De Meirleir L, Lund AM, Gil-Campos M, Van den Hout JMP, Tylki-Szymanska A, Geraci S, Ardigò D, Cattaneo F, Harmatz P, Phillips D. Health Related Quality of Life, Disability, and Pain in Alpha Mannosidosis: Long-Term Data of Enzyme Replacement Therapy With Velmanase Alfa (Human Recombinant Alpha Mannosidase). Journal of Inborn Errors of Metabolism & Screening 2018, Volume 6: 1-12
- [Result] Lund AM, Borgwardt L, Cattaneo F, Ardigo D, Geraci S, Gil-Campos M, De Meirleir L, Laroche C, Dolhem P, Cole D, Tylki-Szymanska A, Lopez-Rodriguez M, Guillen-Navarro E, Dali CI, Heron B, Fogh J, Muschol N, Phillips D, Van den Hout JMH, Jones SA, Amraoui Y, Harmatz P, Guffon N. Comprehensive long-term efficacy and safety of recombinant human alpha-mannosidase (velmanase alfa) treatment in patients with alpha-mannosidosis. J Inherit Metab Dis. 2018 Nov;41(6):1225-1233. doi: 10.1007/s10545-018-0175-2. Epub 2018 May 3. PMID 29725868
- [Result] Harmatz P, Cattaneo F, Ardigo D, Geraci S, Hennermann JB, Guffon N, Lund A, Hendriksz CJ, Borgwardt L. Enzyme replacement therapy with velmanase alfa (human recombinant alpha-mannosidase): Novel global treatment response model and outcomes in patients with alpha-mannosidosis. Mol Genet Metab. 2018 Jun;124(2):152-160. doi: 10.1016/j.ymgme.2018.04.003. Epub 2018 Apr 18. PMID 29716835
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2014-003950-15